CLINICAL TRIAL: NCT02029651
Title: Effects of Novel Game Rehabilitation System (E-glove System) on Upper Extremity Function of Patients With Stroke :Randomized Controlled Trial
Brief Title: Effects of Novel Game Rehabilitation System on Upper Extremity Function of Patients With Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Rehabilitation Center, Seoul, Korea (Other Government)
Collaborators: Ministry of Trade, Industry & Energy, Republic of Korea (Other Government); National IT Industry Promotion Agency, Republic of Korea (Unknown)
Responsible Party: Principal Investigator, Joon-Ho Shin, Manager, National Rehabilitation Center, Seoul, Korea
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NRC-2013-04-035
Record Dates: First submitted 2014-01-01; First posted 2014-01-08 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Stroke
Keywords: Stroke; Hand; Rehabilitation; Game
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- E-glove system (Experimental): E-glove rehabilitation system for upper extremity
  Interventions: Device: E-glove system
- Conventional occupational therapy (Active Comparator): conventional occupational therapy
  Interventions: Procedure: Conventional occupational therapy

INTERVENTIONS:
Device: E-glove system — Novel rehabilitation system using game for upper extremity rehabilitation for patients with stroke
  Arms: E-glove system
Procedure: Conventional occupational therapy — conventional occupational therapy
  Arms: Conventional occupational therapy

SUMMARY:
The purpose of this study is to determine whether novel upper extremity rehabilitation system for patients with stroke(e-glove system) are effective in the rehabilitation compared to conventional occupational therapy

ELIGIBILITY:
Inclusion Criteria:

* Hemiplegic stroke patients
* Medical research council scale >= 2 of finger or wrist flexor/extensor
* Medical research council scale >= 2 of elbow pronation/supination

Exclusion Criteria:

* Bilateral weakness of upper extremities
* Uncontrolled medical or surgical illness
* Predisposing psychological or neurological disorders
* Severe aphasia unable to communicate
* Severe cognitive impairment not to cooperate
* Severe pain impeding upper extremity rehabilitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Fugl-meyer assessment_upper extremity | Change from baseline in Fugl-Meyer assessment at 4 weeks after intervention

SECONDARY OUTCOMES:
Fugl-meyer assessment_upper extremity | Baseline, after 10th intervention, after 20th intervention, 1 month after intervention
Jebsen hand function test | Baseline, after 10th intervention, after 20th intervention, 1 month after intervention
Purdue pegboard | Baseline, after 10th intervention, after 20th intervention, 1 month after intervention
Stroke impact scale | Baseline, after 20th intervention
Modified Ashworth scale of affected upper extremity | Baseline, after 20th intervention
Medical research council scale of muscle strength of affected upper extremity | Baseline,after 20th intervention
Satisfaction about intervention | after 20th intervention
  only for the participants of E-glove intervention

CONTACTS AND LOCATIONS:
Overall Officials: Joon-Ho Shin, Principal Investigator — National Rehabilitation Center
Locations (1):
- National Rehabilitation Center, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Shin JH, Kim MY, Lee JY, Jeon YJ, Kim S, Lee S, Seo B, Choi Y. Effects of virtual reality-based rehabilitation on distal upper extremity function and health-related quality of life: a single-blinded, randomized controlled trial. J Neuroeng Rehabil. 2016 Feb 24;13:17. doi: 10.1186/s12984-016-0125-x. PMID 26911438